CLINICAL TRIAL: NCT00122889
Title: Garlic Metabolism and Cytochrome P450 Modulation
Brief Title: Effects of Garlic Supplements on Drug Metabolism
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Danny Shen, PhD, Fred Hutchinson Cancer Research Center
Other Study IDs: FHCRC-1984.00; R21AT002712-01 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Drug Interactions; Pharmacokinetics; Garlic; Complementary Therapies; Complementary and Alternative Medicine
MeSH Terms: interventions — allyl sulfide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Garlic powder with high allicin content
Drug: Garlic powder with low allicin content
Drug: Garlic oil
Drug: Aged garlic

SUMMARY:
This study will determine whether garlic supplements affect the way certain drugs are processed in the body.

DETAILED DESCRIPTION:
Garlic supplements, which are often used to lower cholesterol and prevent cancer, are one of the most commonly used herbal products in the United States.

However, little is known about the way garlic supplements may interact with prescription medications when used simultaneously. This study will investigate four commonly used garlic supplements: garlic powder with a low content of allicin (a compound with antibacterial properties), garlic powder with a high allicin content, garlic oil, and aged garlic. The effects of these 4 garlic products on the drug-metabolizing enzyme cytochrome P450 (CYP) and a drug transporter, P-glycoprotein (Pgp) will be examined.

Participants will be randomly assigned to receive one of the four garlic supplements for 4 weeks. Drug probes of CYP and Pgp will be used to assess the in vivo activities of the substances. On the first day of garlic ingestion, blood collection will occur immediately after participants ingest their garlic supplement and 3, 4, and 6 hours after ingestion. Urine collection will occur immediately after participants' first garlic ingestion and 12, 15, and 72 hours after ingestion. Blood and urine collection will determine the concentration of the drug probes in the body, which will indicate changes in CYP and Pgp. Blood and urine tests will be repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20 and 32
* Able to read and understand English
* MUST LIVE WITHIN THE SEATTLE, WA AREA.

Exclusion Criteria:

* Current use of herbal medicines other than oral contraceptives
* History of cardiopulmonary, liver, renal or endocrine disease
* Allergy or sensitivity to any of the drugs that will be used in the probe cocktails or the garlic supplements
* Daily consumption of vegetables with a high allium content, including garlic, shallots, leeks, and chives
* Pregnancy or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-07; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Blood plasma and urine samples | 3 months

SECONDARY OUTCOMES:
Blood plasma and breath samples. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Danny D. Shen, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States